CLINICAL TRIAL: NCT01818232
Title: A Phase 1, Open-label, Nonrandomized, Single Dose Study to Evaluate the Absorption, Metabolism, and Excretion of [14C]-LX4211, Following Oral Administration, in Healthy Male Subjects
Brief Title: Study to Determine the Absorption, Metabolism, and Excretion of [14C]LX4211 in Healthy Male Subjects
Acronym: AME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-108-NRM; LX4211.108
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Healthy

ARMS (1):
- [14C]-LX4211 (Experimental): 400 mg LX4211 administered orally
  Interventions: Drug: [14C]-LX4211

INTERVENTIONS:
Drug: [14C]-LX4211

SUMMARY:
This phase 1 study is to evaluate the pharmacokinetics (PK), metabolism, routes and extent of elimination of a single oral dose of 400 mg [14C]LX4211 to healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 to ≤55 years of age
* Vital signs at Screening in the following ranges: systolic blood pressure, 90-140 mm Hg; diastolic blood pressure, 50-90 mm Hg; heart rate, 50-100 bpm
* Body mass index (BMI) ≥18 and ≤35 kg/sq m
* Historically able to produce a minimum of 1 bowel movement per day
* Willing and able to provide written informed consent

Exclusion Criteria:

* Female
* Receipt of any investigational drug within 30 days prior to Dosing, or investigational protein or antibody-based therapeutic agents within 3 months prior to Screening
* Prior exposure to LX4211
* Use any tobacco product within 2 months prior to Screening and while participating in the study (Day -1 through Discharge)
* History of bariatric surgery or any other GI surgery that may induce malabsorption
* History of any major surgery within 6 months prior to Screening
* History of renal or hepatic disease, or significantly abnormal kidney or liver function tests at Screening
* History of any clinically relevant psychiatric, renal, hepatic, pancreatic, cardiovascular, neurological, hematological, or GI abnormality
* History of any active infection within 14 days prior to Dosing
* History of alcohol or substance abuse within 2 years prior to Dosing
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Donation or loss of >400 mL of blood or blood product within 3 months of Dosing
* Positive urine glucose at Screening
* Positive urine screen for drugs of abuse at Screening or Day -1
* Positive breath test for alcohol at Screening or Day -1
* Participation in >1 other radiolabeled investigational study drug trial within 12 months prior to Day -1
* Exposure to significant radiation within 12 months prior to Day -1

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Day 1: predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose

SECONDARY OUTCOMES:
Number of subjects experiencing an adverse event | Day 1 through discharge
Urinary recovery of radioactivity | predose through 24 hours
Fecal recovery of radioactivity | predose through 24 hours
Whole blood and plasma concentration of total radioactivity | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna Ogbaa, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Madison, Wisconsin, United States